CLINICAL TRIAL: NCT07305974
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IIa Clinical Study to Evaluate the Safety, Preliminary Efficacy, and Pharmacokinetic/Pharmacodynamic Characteristics of RG002C0106 Injection in Subjects With Primary IgA Nephropathy
Brief Title: A Phase IIa Clinical Study of RG002C0106 Injection in Subjects With Primary IgA Nephropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rigerna Therapeutics Co., Ltd.; Rigerna Therapeutics (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG002C0106-201
Record Dates: First submitted 2025-12-07; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: IgAN
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: RG002C0106 (Experimental): Randomly enrolled subjects receiving the investigational drug will receive subcutaneous injection for administration
  Interventions: Drug: RG002C0106
- Placebo Comparator: placebo (Placebo Comparator): Randomly enrolled subjects receiving placebo will receive subcutaneous injection for administration
  Interventions: Drug: placebo subcutaneous administration

INTERVENTIONS:
Drug: RG002C0106 — RG002C0106 for subcutaneous (SC) injection
  Arms: Experimental: RG002C0106
Drug: placebo subcutaneous administration — The placebo is made of normal saline.
  Arms: Placebo Comparator: placebo

SUMMARY:
This study looks at how well and safely RG002C0106 works for patients with certain kidney disease: primary IgA nephropathy. It's a phase IIa trial done at several locations where both patients and doctors unknow what treatment is being given.

DETAILED DESCRIPTION:
This is a Phase IIa, multicenter, double-blind clinical trial designed to evaluate the efficacy and safety of RG002C0106 in patients with primary IgA nephropathy. The primary objective is to assess the efficacy of RG002C0106 in reducing urinary protein excretion and preserving renal function in these patients. Secondary objectives include characterization of the safety profile, pharmacokinetics, and pharmacodynamics of the treatment

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial and sign the informed consent form (ICF);
2. Male or female participants aged 18 to 65 years (inclusive) at the time of signing the ICF;
3. Body weight ≥ 40 kg;
4. Negative blood pregnancy test result at screening for female participants of childbearing potential;
5. Renal biopsy pathology results within 10 years prior to screening confirming a diagnosis of primary IgA nephropathy;
6. 24-hour urinary protein ≥ 0.75 g/24 h during the screening period;
7. Estimated glomerular filtration rate (eGFR) (calculated using the creatinine-based CKD-EPI formula) ≥ 30 mL/min/1.73 m² during the screening period;
8. Must have received vaccination against Neisseria meningitidis (serogroups A, C, W, Y) and Streptococcus pneumoniae infections at least 2 weeks prior to the first dose of the investigational product and provide proof of such vaccination;
9. Participants must agree and require their partners to use adequate contraception from the time of signing the ICF, throughout the study, and for at least 3 months after the study ends . Male participants must not donate sperm for at least 6 months after the last dose of the investigational product.

Exclusion Criteria:

1. Patients with secondary IgA nephropathy ;
2. Renal biopsy pathology shows renal tubular atrophy or interstitial fibrosis ≥ 50%; or crescent formation in ≥ 50% of glomeruli ;
3. Acute kidney injury or rapidly progressive glomerulonephritis within 4 weeks prior to screening ;
4. Patients with nephrotic syndrome, defined as: 24-hour urinary protein (24h-UP) >3.5 g with hypoalbuminemia (serum albumin <3.0 g/dL), hypercholesterolemia (total cholesterol >350 mg/dL), and edema;
5. Any of the following abnormal laboratory results at screening:

   * Alanine aminotransferase (ALT) > 2 × upper limit of normal (ULN);
   * Total bilirubin (TB) > 1.5 × ULN. However, for patients with a confirmed diagnosis of Gilbert's syndrome, if TB > 1.5 × ULN but conjugated bilirubin < ULN, they may be enrolled;
6. Positive test results at screening for HBsAg, HCV Ab,HIV-IgG, or TP-Ab;
7. Poorly controlled type 1 or type 2 diabetes during the screening period ;
8. Persistent clinically significant elevated blood pressure during the screening period ;
9. Patients with immunodeficiency diseases;
10. Patients with splenic insufficiency (e.g., asplenia or history of splenectomy);
11. History of kidney transplantation or organ transplantation (including bone marrow transplantation, stem cell transplantation, etc.);
12. Suspected or confirmed history of hereditary complement deficiency;
13. History of any tumor within 5 years before screening, except for the following: basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, and squamous cell carcinoma of the skin that have been completely cured after treatment;
14. History of meningococcal infection within 12 months before screening;
15. Active or suspected viral, bacterial, fungal, or parasitic infection within 14 days prior to investigational product administration;
16. History of allergic reactions to oligonucleotides or N-acetylgalactosamine (GalNAc);
17. History of intolerance to subcutaneous injections or significant abdominal scarring that may impede administration or local tolerance assessment of the investigational product;
18. Treatment with small-molecule complement inhibitors (e.g., iptacopan) within 3 months prior to investigational product administration, or previous treatment failure or intolerance;
19. History of clinically significant severe infection within 3 months prior to screening, as determined by the investigator;
20. Major surgery or severe trauma within 3 months prior to investigational product administration, incomplete recovery, or planned surgery during the study;
21. Participation in any investigational drug or medical device clinical trial within 1 month prior to investigational product administration (excluding screen failures);
22. Any other condition considered by the investigator to make the participant unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
The percentage change from baseline in the mean 24hUPCR)at Week 24 after the first subcutaneous admini; | up to 169 days
Incidence of adverse events (AEs) and serious adverse events (SAEs) related to the investigational drug. | up to 169 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No